CLINICAL TRIAL: NCT07080372
Title: Role of Early Arterial Phase Imaging in Accurately Differentiating Hepatocellular Carcinoma From Dysplastic Nodules in Cirrhotic Patients
Brief Title: Role of Early API in Accurately Differentiating Hepatocellular Carcinoma From Dysplastic Nodules in Cirrhotic Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/926
Record Dates: First submitted 2025-06-28; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Dysplastic Nodule

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: assesment — This study aims to assess the role of early arterial phase in detecting and differentiating hepatocellular carcinoma from dysplastic nodules in chronic liver disease patients.

SUMMARY:
Liver cirrhosis is a common consequence of chronic liver disease, resulting from sustained hepatic injury due to various etiologies. Cirrhosis predisposes individuals to the development of hepatocellular carcinoma (HCC), the most prevalent primary malignancy of the liver. Among cirrhotic patients, distinguishing between hepatocellular carcinoma and dysplastic nodules is crucial for timely diagnosis, treatment planning, and prognostic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with abnormal LFTs
* Liver lesions of various sizes
* Patients with chronic liver disease
* Individuals undergoing routine liver screening
* Willing participants who consent to the study

Exclusion Criteria:

* Children less than 5years
* Patients who are allergic or have a history of allergy to contrast media
* Patients with deranged renal function tests
* Pregnant women

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Aim of the study: This study aims to assess the role of early arterial phase in detecting and differentiating hepatocellular carcinoma from dysplastic nodules in chronic liver disease patients
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
self administered proforma form | 12 Months
  A clinical history form is a structured document used to gather comprehensive information about a patient's medical background and current health status. It typically includes sections for identifying patient demographics, past medical history, family history, social history, medications, allergies, and a detailed account of the current illness or complaint.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore General Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No